CLINICAL TRIAL: NCT02603744
Title: Evaluate the Safety and Feasibility of Intra-ovarian Injection of Autologous Adipose Derived Mesenchymal Stromal Cells (ADMSC) in Women With Premature Ovarian Failure(POF)
Brief Title: Autologous Adipose Derived Mesenchymal Stromal Cells Transplantation in Women With Premature Ovarian Failure (POF)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rep-Bio-Royan-001
Record Dates: First submitted 2015-11-07; First posted 2015-11-13 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Premature Ovarian Failure
Keywords: Premature ovarian failure adipose derived stromal cells intraovarian injection
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5 million MSC (Experimental): The patients with POF who underwent intraovarian injection of 5 million mesenchymal stem cells.
  Interventions: Biological: Intraovarian injection of Adipose derived Stromal cells (ADSCs)
- 10 million MSC (Experimental): The patients with POF who underwent intraovarian injection of 10 million mesenchymal stem cells.
  Interventions: Biological: Intraovarian injection of Adipose derived Stromal cells (ADSCs)
- 15 million MSC (Experimental): The patients with POF who underwent intraovarian injection of 15 million mesenchymal stem cells.
  Interventions: Biological: Intraovarian injection of Adipose derived Stromal cells (ADSCs)

INTERVENTIONS:
Biological: Intraovarian injection of Adipose derived Stromal cells (ADSCs) — Intra-ovarian injection of Adipose derived mesenchymal stem cells.
  Other Names: stem cell transplantation

SUMMARY:
The goal of this study is to determine safety and tolerability and of intra-ovarian injection of adipose derived stromal cell in women with premature ovarian failure and to study the preliminary efficacy ADSCs intra ovarian injection on ovarian function improvement.

DETAILED DESCRIPTION:
In this study 9 patients with the diagnosis of premature ovarian failure will participate.

The patients will be divided randomly in 3 groups, each group contains 3 patients. First group will receive 5 millions of ADSCs, second group receive 10 millions cells and the third group receive 15millions of ADSCs.

Stem cell Transplantation method is intraovarian injection of ADSCs which will be performed under guidance of transvaginal sonography.

All the patients will be followed for 12 months after cell injection to evaluate any adverse events .

ELIGIBILITY:
Inclusion Criteria:

* female
* Age : 20-39
* FSH>20

Exclusion Criteria:

* liposuction contraindication
* thyroid dysfunction
* immune system disease
* past history of cancer , chemotherapy , radiotherapy
* HIV+, hepatitis B, C
* Severe endometriosis

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
ovary mass | up to 12months
  Evaluation the formation of ovary mass by sonography up to one year after transplantation (patient will follow for any adverse event via follow up visits (24hr after transplantation, 1th , 2th , 4th , 8th , 12th week , 6th month and 12th month after cell transplantation.
ovary abcess | Up to 12 months
  Evaluation the ovary abcess formation up to one year after transplantation (patient will follow for any adverse event via follow up visits (24hr after transplantation, 1th , 2th , 4th , 8th , 12th week , 6th month and 12th month after cell transplantation.

SECONDARY OUTCOMES:
Follicle Stimulating Hormone (FSH) serum level | Up to 12months
  one year after transplantation (patient will follow for any adverse event via one year after transplantation ( this measures will evaluate within follow up visits at 1th , 2th , 4th, 8th, 12th weeks and 6th and 12th month after transplantation
Anti-Mullerian Hormone (AMH) serum level | Up to 12months
  Evaluation the AMH serum level by blood sampling up to one year after transplantation (patient will follow for any adverse event via one year after transplantation ( this measures will evaluate within follow up visits at 1th , 2th , 4th, 8th, 12th weeks and 6th and 12th month after transplantation
Number of antral follicle | Up to 12months
  Evaluation the number of antral follicle by sonography up to one year after transplantation ( this measures will evaluate within follow up visits at 1th , 2th , 4th, 8th, 12th weeks and 6th and 12th month after transplantation
Antral follicle volume | Up to 12months
  Evaluation the antral follicle volume by sonography up to one year after transplantation ( this measures will evaluate within follow up visits at 1th , 2th , 4th, 8th, 12th weeks and 6th and 12th month after transplantation
Menstruation recurrence rate | Up to 12 months
  Evaluation the menstruation recurrence rate up to one year after transplantation ( this measures will evaluate within follow up visits at 1th , 2th , 4th, 8th, 12th weeks and 6th and 12th month after transplantation
Pregnancy rate | Up to 12months
  Evaluation the pregnancy rate up to one year after transplantation ( this measures will evaluate within follow up visits at 1th , 2th , 4th, 8th, 12th weeks and 6th and 12th month after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Tahereh Madani, MD, Study Director — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Mehri Mashayekhi, MD, Study Director — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Elham sadat Mirzadeh, MD, Principal Investigator — Department of Regenerative Medicin, Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Mashayekhi M, Mirzadeh E, Chekini Z, Ahmadi F, Eftekhari-Yazdi P, Vesali S, Madani T, Aghdami N. Evaluation of safety, feasibility and efficacy of intra-ovarian transplantation of autologous adipose derived mesenchymal stromal cells in idiopathic premature ovarian failure patients: non-randomized clinical trial, phase I, first in human. J Ovarian Res. 2021 Jan 6;14(1):5. doi: 10.1186/s13048-020-00743-3. PMID 33407794
- See also: Related Info — http://RoyanInstitute.org